CLINICAL TRIAL: NCT06966999
Title: Efficacy of Botulinum Toxin Type A for Acute Acquired Comitant Esotropia: An Age-Stratified Two-Year Follow-Up Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-073
Record Dates: First submitted 2025-04-28; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-04

CONDITIONS: Acute Acquired Comitant Esotropia
Keywords: Botulinum toxin; esotropia
MeSH Terms: conditions — Esotropia | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- To assess and compare the long-term efficacy of botulinum toxin type A （BTXA) in the treatment of ac (Other)
  Interventions: Procedure: Botulinum Toxin Type A Injection [Botox]

INTERVENTIONS:
Procedure: Botulinum Toxin Type A Injection [Botox] — for patients >12 years presenting with large-angle esotropia (>50 PD), primary surgical intervention was recommended as the preferred approach to minimize failure and recurrence risk. Conversely, for patients ≤12 years, BTXA injection was maintained as the first-line treatment regardless of the deviation angle.

SUMMARY:
The goal of this clinical trial is to assess and compare the efficacy of two-year follow-up botulinum toxin type A （BTXA) in the treatment of acute acquired comitant esotropia (AACE) across five age groups: ≤6 years, >6 to ≤12 years, >12 to ≤20 years, >20 to ≤30 years, and >30 years. For patients >12 years presenting with large-angle esotropia (>50 PD), primary surgical intervention was recommended as the preferred approach to minimize failure and recurrence risk. Conversely, for patients ≤12 years, BTXA injection was maintained as the first-line treatment regardless of the deviation angle.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute acquired comitant esotropia (AACE) with sudden onset and diplopia
* Normal eye movements with deviation difference ≤5 prism diopters (PD) in all gaze directions
* Hyperopia < +3.00 diopters
* <10 PD reduction in esotropia with hypermetropic spectacle correction
* No prior extraocular muscle surgery
* Absence of congenital/developmental anomalies affecting treatment outcomes

Exclusion Criteria:

* Deviation difference >5 PD in any gaze direction
* Hyperopia ≥ +3.00 diopters
* History of extraocular muscle surgery
* Presence of congenital/developmental anomalies potentially impacting outcomes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
the cumulative motor success rate | 2 years
  Kaplan-Meier survival analyses were conducted to evaluate the cumulative motor success rate.
  A successful motor outcome was defined as achieving orthotropic alignment within 8 PD at both near (33 cm) and distance (6 m) fixation, accompanied by complete resolution of diplopia.

SECONDARY OUTCOMES:
the sensory success rate | 2 years
  The sensory success rate was calculated as the proportion of patients achieving successful sensory outcomes among all AACE patients receiving BTXA treatment, expressed as:
  Sensory success rate = (Number of AACE patients with successful sensory outcomes post-BTXA) / (Total number of AACE patients treated with BTXA) × 100% Sensory success was defined as the restoration of stereopsis.

OTHER OUTCOMES:
the hazard ratio (HR) for the risk of AACE relapse | 2 years
  AACE relapse was identified by either the recurrence of diplopic symptoms or the re-emergence of esotropia >8 PD. The Cox proportional hazards model was used to identify potential risk factors for AACE relapse.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China